CLINICAL TRIAL: NCT04011943
Title: Study of the Effects of Fecal Microbiota Transplantation for Correction of the Physiological State of the Human Body in Norm and in Pathology
Brief Title: Fecal Microbiota Transplantation for Health Improvement (TFM3)
Acronym: TFM3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal Research and Clinical Center of Physical-Chemical Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFM3
Record Dates: First submitted 2019-05-17; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Ulcerative Colitis; Irritable Bowel Syndrome; Crohn Disease; Irritable Bowel
MeSH Terms: conditions — Colitis, Ulcerative; Irritable Bowel Syndrome; Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: In total, 85 participants must be registered. 35 are healthy volunteers. Of these volunteers, 15 will receive autologous transplantation of fecal microbiota, 10 will receive both autologous and heterologous transplantation and 10 volunteers form a placebo-controlled group.
  50 participants will form a treatment group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants with bowel diseases (Experimental): Treatment by transplantation of fecal microbiota
  Interventions: Other: Fecal Microbiota Transplantation
- autologous transplantation of fecal microbiota - healthy (Experimental): Healthy volunteers will receive autologous transplantation of fecal microbiota (capsules)
  Interventions: Other: Fecal Microbiota Transplantation
- Both autologous and heterologous transplantation - healthy (Experimental): Healthy volunteers will receive both autologous and heterologous transplantation (capsules)
  Interventions: Other: Fecal Microbiota Transplantation
- placebo capsules - healthy (Placebo Comparator): Healthy volunteers will receive placebo capsules
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation

SUMMARY:
Search for mechanisms of the effect of fecal transplantation on a healthy organism and various nosological forms.

DETAILED DESCRIPTION:
Objectives of the study:

1. To select donors of fecal samples for carrying out the procedure of fecal transplantation of microbiota to patients with various nosological forms.
2. To select healthy volunteers for autologous and heterologous transfusion of feces and a group of placebo-control.
3. Create a bank of fecal samples of healthy donors;
4. Conduct a procedure for fecal microbiota transplantation for a sample of patients and healthy volunteers;
5. Analyze the efficacy of therapy with TFM on the sample of patients;
6. Analyze the effect of autologous, heterologous TFM and placebo on healthy volunteers;
7. Analyze long-term effects in patients within 6 months after the TPM.

The study is expected to include 50 patients, 35 healthy volunteers and healthy feces donors The study is scheduled to begin in May 2018, the supposed completion of the study is December 2020

ELIGIBILITY:
Inclusion Criteria:

* the age of patients - from 18 to 75 years, both sexes;
* Patients with:

  * antibiotic-associated colitis,
  * inflammatory bowel diseases (ulcerative colitis, Crohn's disease),
  * diseases caused by C. difficile infection,
  * a syndrome of impaired intestinal absorption,
  * irritable bowel syndrome,
  * celiac disease (severe form),
  * metabolic syndrome, including diabetes mellitus type II,
  * Atopic dermatitis with damage to the mucous membrane of the colon,
  * hepatitis of various etiologies,
  * cirrhosis of the liver of various etiologies
  * pancreatitis of various etiologies,
* Absence of contraindications to gastroscopy
* informed consent of the patient for the transplant procedure

Exclusion Criteria:

* the presence of a concomitant chronic infectious or neoplastic disease in the patient
* Patients with a proven allergy to foods not excluded from the donor's diet
* absence of the patient for one or more intermediate stages of the examination.
* informed refusal to continue therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Ulcerative Colitis remission | 1 month after transplantation. Change from Baseline - 1 day before transplantation
  Ulcerative Colitis remission defined as a Simple Clinical Colitis Activity Index <3
Crohn Disease remission | 1 month after transplantation. Change from Baseline - 1 day before transplantation.
  Crohn Disease remission defined as a Harvey-bradshaw index <3.

SECONDARY OUTCOMES:
Improvement in Ulcerative Colitis symptoms. | 1 month after transplantation. Change from Baseline - 1 day before transplantation.
  Defined as improvement in SCCAI.
Change in gut microbiome | 1 month after transplantation. Change from Baseline - 1 day before transplantation.
  Diversity and variability of gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ilina, MD, Principal Investigator — FRCC PCM
Locations (1):
- FRCC PCM, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No